CLINICAL TRIAL: NCT05126459
Title: A Comparison of Oral Sedation-related Events of Three Multiagent Oral Sedation Regimens in Pediatric Dental Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Jung-Wei Chen, DDS, MS, PhD, Program Director, Pediatric Dentistry, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5190213
Record Dates: First submitted 2021-11-08; First posted 2021-11-19 (Actual); Results first posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Anxiety, Dental; Dental Decay
Keywords: Pediatric; Dental
MeSH Terms: conditions — Anxiety Disorders; Dental Caries | interventions — ICE protocol 3

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Regimen 1 (Active Comparator): Oral administration - Hydroxyzine (1.5 - 2mg/kg) Oral administration - Meperidine (1.5 -2 mg/kg) Oral administration - Midazolam (0.5- 0.75 mg/kg) Inhalation - Nitrous oxide/oxygen (30-50% N2O/ 70-50% O2)
  Interventions: Combination Product: Regimen 1
- Regimen 2 (Experimental): Oral administration - Hydroxyzine (1.5 - 2mg/kg) Oral administration- Meperidine (1.5 -2 mg/kg) Inhalation - Nitrous oxide/oxygen (30-50% N2O/ 70-50% O2) -
  Interventions: Combination Product: Regimen #2
- Regimen 3 (Experimental): Oral administration - Hydroxyzine (1.5 - 2mg/kg) Oral administration - Midazolam (0.5- 0.75 mg/kg) Inhalation- Nitrous oxide/oxygen (30-50% N2O/ 70-50% O2)
  Interventions: Combination Product: Regimen #3

INTERVENTIONS:
Combination Product: Regimen 1 — Administer orally after informed consent obtained prior to any dental procedure. Hydroxyzine (1.5- 2mg/kg) + Meperidine (1.5 -2 mg/kg) + Midazolam (0.5- 0.75 mg/kg) In combination with oral drugs stated above, administeration via inhalation of Nitrous oxide/oxygen (30-50% N2O/ 70-50% O2) via inhalation.
  Arms: Regimen 1
Combination Product: Regimen #2 — Administer orally after informed consent obtained prior to any dental procedure. Hydroxyzine (1.5 - 2mg/kg) + Meperidine (1.5 -2 mg/kg). Administer Nitrous oxide/oxygen (30-50% N2O/ 70-50% O2) via inhalation.
  Arms: Regimen 2
Combination Product: Regimen #3 — Administer orally after informed consent obtained prior to any dental procedure. Hydroxyzine (1.5 - 2mg/kg) + Midazolam (0.5- 0.75 mg/kg). Administer Nitrous oxide/oxygen (30-50% N2O/ 70-50% O2) via inhalation.
  Arms: Regimen 3

SUMMARY:
This study will compare the post sedation events from three different multi-drug oral sedation regimens in order to help pediatric dentists determine the best course of action for their patients and prepare parents appropriately and caution them about the expected effects. Patients will be evaluated for adverse effects within two time periods at 8 and 24 hours post oral sedation procedure using surveys.

DETAILED DESCRIPTION:
Inclusion criteria included patients of record who were scheduled to undergo oral sedation at Loma Linda University Pediatric Dentistry clinic for dental treatment. Children ages ranged from 3 to 6 years old with no medical issues, ASA-1. The reason for oral sedation was situational anxiety in the dental operatory. Exclusion criteria included children who presented with a history of: (1) acute illness; (2) upper respiratory tract infection within two weeks of treatment; (3) taking any medication within the two weeks prior to scheduled dental treatment; and (4) a body mass index (BMI) greater than the 95th percentile for their age and gender. A total sample of 60 healthy pediatric patients were included in this study with were no gender, race, or ethnic significant difference.

The included patients were randomly allocated into one of three sedation groups by drawing a concealed folded paper from an opaque randomization bag after obtaining parent consent. All papers that were used in the randomization had the same size and texture. The pediatric dental resident and attending faculty were informed with medication combination once randomized allocation had been made.

The study groups were as follows: Group 1 received Midazolam (0.5- 0.75 mg/kg), Meperidine (1.5-2.0 mg/kg), and Hydroxyzine (1.5- 2.0 mg/kg), Group 2 received Meperidine (1.5-2 mg/kg) and Hydroxyzine (1.5- 2.0 mg/kg). Group 3 received Midazolam (0.5- 0.75 mg/kg) and Hydroxyzine (1.5- 2mg/kg).

Clinical Procedure Calculations based on the child's weight of maximum local anesthetic delivery, oral sedation medication dosages, and reversal agents were completed prior to delivery of medication. The reversal agent used for benzodiazepines was Flumazenil, 0.01mg/Kg with a maximum of 0.2 mg/dose. While the reversal agent for Meperidine was Naloxone, calculated as 0.1 mg/Kg up to 2 mg.

After obtaining proper consents, all patients were placed in passive protective stabilization (Joey Board®, Joey Board, Queen Creek, AZ) in the event the child was to become uncooperative and to maintain patient stability during treatment, as coordination could be impaired. Nitrous oxide/Oxygen (N2O/O2) was used in all sedations and administered at a flow rate of four to six L/minute (30-50% N2O/ 10-50% O2) with 100% O2 given for five minutes pre- and postoperatively. All operating dentists followed standard sedation protocol at standard sedation protocol in Loma Linda University Pediatric Dentistry Clinic adapted from the American Academy of Pediatric Dentistry (AAPD) guidelines.8 Routine dental care was provided with local anesthesia with rubber dam or isolite® isolation. Xylocaine (2% lidocaine with 1:100,000 epinephrine) was used for local anesthesia in all cases and did not exceed 4 mg/kg lidocaine. Once AAPD discharge criteria8 were met, the patient was released to the parent. At that time, postoperative care instructions, including emergency contact numbers and recommendation for over-the-counter pain medications, if needed, were provided both verbally and in written form.

The dentist performing each sedation was asked to complete a detailed questionnaire that provided details about the patient's behavior from the time of drug administration to the time of discharge (Survey 1). In addition, parents received two telephone interviews regarding events that occurred after the sedation session. An investigator conducted all phone interviews. These phone interviews took place at eight hours (Survey 2) and 24 hours (Survey 3) after discharge.

For all three of the surveys, questions were designed to elucidate patient physical signs and/or behaviors that fell into the following categories: (1) sleep disturbances; (2) gastrointestinal side effects; (3) non-aggressive behavior changes; (4) residual central nervous system alterations; (5) respiratory depression; (6) musculoskeletal effects; (7) physical reactions; (8) existence of a paradoxical reaction; and (9) amnesic effects. Information on the pre-sedation cooperation level and overall effectiveness of the sedation (rated as ineffective, effective, very effective, or overly sedated) were obtained from the procedural sedation record (adopted from AAPD) corresponding to each case.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo oral sedation appointments in Loma Linda University Pediatric dental clinic for operative procedures.
* Age 3-7 years old, Healthy ( ASA-1 )
* No gender, race or ethnic restrictions.
* Reason for conscious oral sedation is situational anxiety in the dental operatory

Exclusion Criteria:

* Children with a history of acute illness
* History upper respiratory tract infection within two weeks of treatment
* Children taking any medication within the two weeks prior to scheduled dental treatment
* Sedation within the last six months
* Body mass index (BMI) greater than the 95th percentile for their age and sex
* Failing to drink the entire amount of sedation medications dispensed

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Wei Chen, DDS,MS,PhD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Regimen 1 | Regimen 2 | Regimen 3
Started | 20 | 20 | 20
Completed | 20 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: pediatric dental patient with situational anxiety in dental operatory settings.
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen 1 | Regimen 2 | Regimen 3 | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Customized [Mean (Standard Deviation); unit: Month]
  Age, month | 65.25 (13.09) | 65.10 (11.87) | 60.30 (12.2) | 63.55 (12.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 9 | 35
  Male | 5 | 9 | 11 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Sedation-Related Events in Musculoskeletal System During Sedation
Description: Compare the incidence of adverse sedation related events (categories: amount and frequency of sleeping, level of activity, gastrointestinal discomfort, central nervous system, respiratory depression, paradoxical reactions) between three different multi-agent oral sedation regimens in LLUSD pediatric dental patients who were scheduled for oral sedation.
  Data will be collected in the form of 3 survey sets: the surveys is survey set 1 are written surveys to be completed by the dentist (Survey 1), and survey sets 2&3 are phone surveys to be conducted by the researcher with the parents 8 (eight) hours (Survey 2) and 24 (twenty-four) hours (Survey 3) after discharge Musculoskeletal system reaction during sedation scale: This is the result for Musculoskeletal related questions, it is a sum of 3 yes or no questions. (minimum=0, maximum=3) The higher the worse.
Time Frame: during sedation
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Regimen 1 | Regimen 2 | Regimen 3
Number analyzed (Participants) | 20 | 20 | 20
score on a scale | 2.8 [2.67 to 3] | 3 [3 to 3] | 2.5500 [2.2 to 2.9]
Statistical Analysis 1: Comparison: Regimen 1 vs Regimen 2 vs Regimen 3; Null hypothesis: there is no significant difference in Musculo skeletal related sedation related events during sedation; Test type: Superiority; p = 0.016, ANOVA — The threshold for statistical significance was p=0.05

2. Primary Outcome: Incidence of Adverse Sedation-Related Events in Musculoskeletal in 8 Hours
Description: Compare the incidence of adverse sedation related events (categories: amount and frequency of sleeping, level of activity, gastrointestinal discomfort, central nervous system, respiratory depression, paradoxical reactions) between three different multi-agent oral sedation regimens in LLUSD pediatric dental patients who were scheduled for oral sedation.
  Data will be collected in the form of 3 survey sets: the surveys is survey set 1 are written surveys to be completed by the dentist (Survey 1), and survey sets 2&3 are phone surveys to be conducted by the researcher with the parents 8 (eight) hours (Survey 2) and 24 (twenty-four) hours (Survey 3) after discharge.
  Musculoskeletal system reaction at 8 hours scale: This is the result for Musculoskeletal related questions, it is a sum of 2 yes or no questions. (minimum=0, maximum=2) The higher the worse.
Time Frame: Change 8 (eight) hours post oral sedation medication administration
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Regimen 1 | Regimen 2 | Regimen 3
Number analyzed (Participants) | 20 | 20 | 20
score on a scale | 0.5 [0.11 to 0.88] | 0.2 [0.007 to 0.39] | 0.2 [0.044 to 0.44]
Statistical Analysis 1: Comparison: Regimen 1 vs Regimen 2; Null hypothesis: there is no significant difference in Musculo skeletal related sedation related events at 8 hours after sedation; Test type: Superiority; p = 0.211, ANOVA — The threshold for statistical significance was p=0.05

3. Primary Outcome: Incidence of Adverse Sedation-Related Events in Musculoskeletal at 24 Hours After Sedation
Description: Compare the incidence of adverse sedation related events (categories: amount and frequency of sleeping, level of activity, gastrointestinal discomfort, central nervous system, respiratory depression, paradoxical reactions) between three different multi-agent oral sedation regimens in LLUSD pediatric dental patients who were scheduled for oral sedation.
  Data will be collected in the form of 3 survey sets: the surveys is survey set 1 are written surveys to be completed by the dentist (Survey 1), and survey sets 2&3 are phone surveys to be conducted by the researcher with the parents 8 (eight) hours (Survey 2) and 24 (twenty-four) hours (Survey 3) after discharge.
  Musculoskeletal system reaction at 24 hours scale: This is the result for Musculoskeletal related questions, it is a sum of 2 yes or no questions. (minimum=0, maximum=2) The higher the worse.
Time Frame: Change between 24 (twenty-four) hours post oral sedation
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Regimen 1 | Regimen 2 | Regimen 3
Number analyzed (Participants) | 20 | 20 | 20
score on a scale | 0.05 [0.005 to 0.15] | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Regimen 1 vs Regimen 2 vs Regimen 3; Test type: Superiority; p = 0.374, ANOVA — The threshold for statistical significance was p=0.05

4. Primary Outcome: Compare Incidence of Adverse Effect Related to Gastrointestinal Reaction During Sedation
Description: Compare the number and type of adverse effect related gastrointestinal reactions.
  Data will be collected in the form of 3 survey sets: the surveys is survey set 1 are written surveys to be completed by the dentist (Survey 1), and survey sets 2&3 are phone surveys to be conducted by the researcher with the parents 8 (eight) hours (Survey 2) and 24 (twenty-four) hours (Survey 3) after discharge.
  GI effect for during sedation score; This is a summary of 3 yes/no questions, Minimum = 0 Maximum =3, the higher means more GI reactions, the worse outcome
Time Frame: During sedation
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Regimen 1: Regimen 1: Administer orally after informed consent obtained prior to any dental procedure. Hydroxyzine (1.5- 2mg/kg) + Meperidine (1.5 -2 mg/kg) + Midazolam (0.5- 0.75 mg/kg) In combination with oral drugs stated above, administration via inhalation of Nitrous oxide/oxygen (30-50% N2O/ 70-50% O2) via inhalation.
Arm/Group | Regimen 1 | Regimen 2 | Regimen 3
Number analyzed (Participants) | 20 | 20 | 20
score on a scale | 0.1 [0.10 to 0.30] | 0.05 [0.05 to 0.15] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Regimen 1 vs Regimen 2 vs Regimen 3; Null hypothesis: there is no significant difference in GI reaction between the 3 regimens; Test type: Superiority; p = 0.55, ANOVA

5. Primary Outcome: Compare Incidence of Adverse Effect Related to Gastrointestinal Reaction 8 Hours After Sedation
Description: Compare the number and type of adverse effect related gastrointestinal reactions Data will be collected in the form of 3 survey sets: the surveys is survey set 1 are written surveys to be completed by the dentist (Survey 1), and survey sets 2&3 are phone surveys to be conducted by the researcher with the parents 8 (eight) hours (Survey 2) and 24 (twenty four) hours (Survey 3) after discharge.
  GI effect 8 hours after sedation score; This is a summary of 5 yes/no questions, Minimum = 0 Maximum =5, the higher means more GI reactions, the worse outcome.
Time Frame: 8 hours after sedation
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | Regimen 1 | Regimen 2 | Regimen 3
Number analyzed (Participants) | 20 | 20 | 20
score on a scale | 0.25 [0.08 to 0.58] | 0 [0 to 0] | 0.05 [0.05 to 0.15]
Statistical Analysis 1: Comparison: Regimen 1 vs Regimen 2 vs Regimen 3; Null hypothesis: there is no significant difference in GI reaction between the 3 regimens 8 hours after sedation; Test type: Superiority; p = 0.16, ANOVA — The threshold for statistical significance was p=0.05

6. Primary Outcome: Compare Incidence of Adverse Effect Related to Gastrointestinal Reaction 24 Hours After Sedation
Description: Compare the number and type of adverse effect related gastrointestinal reactions Data will be collected in the form of 3 survey sets: the surveys is survey set 1 are written surveys to be completed by the dentist (Survey 1), and survey sets 2&3 are phone surveys to be conducted by the researcher with the parents 8 (eight) hours (Survey 2) and 24 (twenty four) hours (Survey 3) after discharge.
  Long term effect for 24 hours after sedation score; This is a summary of 5 yes/no questions, Minimum = 0 Maximum =5, the higher means more GI reactions, the worse outcome
Time Frame: 24 hours after sedation
Measure: Mean (90% Confidence Interval); unit: score on a scale
Arm/Group | Regimen 1 | Regimen 2 | Regimen 3
Number analyzed (Participants) | 20 | 20 | 20
score on a scale | 0.2 [0.007 to 0.39] | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Regimen 1 vs Regimen 2 vs Regimen 3; Null hypothesis: there is no significant difference in GI reaction between the 3 regimens at 24 hours after sedation; Test type: Superiority; p = 0.012, ANOVA — The threshold for statistical significance was p=0.05

ADVERSE EVENTS:
Time Frame: Up to 48 hours post sedation
Description: Delayed communication with some parents, up to 48 hours post sedation.
Arm/Group | Regimen 1 | Regimen 2 | Regimen 3
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 7/20 | 1/20 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen 1 (N=20) | Regimen 2 (N=20) | Regimen 3 (N=20)
Sleep Disturbance (Nervous system disorders) | 1 | 0 | 0 — Bad dreams
Non-Aggressive Behavioral Changes (Nervous system disorders) | 1 | 0 | 1
Gastrointestinal Upset (Gastrointestinal disorders) | 1 | 0 | 0 — Diarrhea Constipation
Respiratory Effects (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 — Snore, difficult to awaken.
Musculoskeletal Effects (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Paradoxical Effects (Nervous system disorders) | 1 | 1 | 0 — Hyperactive

LIMITATIONS AND CAVEATS:
The dentists providing sedation were trained to evaluate behavior parameters, but there may have been difficulty in quantifying parameters due to experience and assessment subjectivity.

All dental treatment was performed with physical stabilization devices, which may have potentially altered the ability to evaluate some of the patients' responses. The postoperative phone calls proved challenging due to difficulty reaching the guardians within the 24 hour phone call window period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/59/NCT05126459/Prot_SAP_002.pdf
  • Informed Consent Form (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/59/NCT05126459/ICF_003.pdf